CLINICAL TRIAL: NCT01605084
Title: An Open-Label Phase 3B Study in HIV-Infected Individuals With Viremia on or After Their First-Line Non-Nucleoside Reverse Transcriptase Inhibitor or Integrase Inhibitor-Based Regimen and Starting a Second-Line Regimen Consisting of ATV/RTV or DRV/RTV With an Optimized NRTI Backbone
Brief Title: Second-line Treatment of HIV-1 With Ritonavir Boosted Atazanavir or Darunavir With an Optimized NRTI Backbone
Acronym: SUPPRESS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI424-493; 2011-006186-18 (EudraCT Number)
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: HIV
MeSH Terms: interventions — Atazanavir Sulfate; Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: ATV/RTV 300/100 mg QD + optimized NRTI backbone (Experimental)
  Interventions: Drug: Atazanavir; Drug: Ritonavir; Drug: Optimized NRTI backbone
- Arm 2: DRV/RTV 800/100 mg QD + optimized NRTI backbone (Experimental)
  Interventions: Drug: Darunavir; Drug: Ritonavir; Drug: Optimized NRTI backbone

INTERVENTIONS:
Drug: Atazanavir — Capsule, Oral, 300 mg, Once daily (QD), 48 weeks
  Other Names: REYATAZ®
  Arms: Arm 1: ATV/RTV 300/100 mg QD + optimized NRTI backbone
Drug: Darunavir — Oral, Two 400 mg Tablets, Once daily (QD), 48 weeks
  Other Names: PREZISTA®
  Arms: Arm 2: DRV/RTV 800/100 mg QD + optimized NRTI backbone
Drug: Ritonavir — Tablet, Oral, 100 mg, Once daily (QD), 48 weeks
  Other Names: NORVIR®
Drug: Optimized NRTI backbone — tablet/capsule, Noninvestigational products i.e. NRTI backbone will be administered according to their respective package inserts for 48 weeks
  NRTI backbone are:
  - Abacavir (300 mg), Tenofovir (300 mg), Didanosine (250 mg or 400 mg), Stavudine (30 mg or 40 mg), Emtricitabine (200 mg), Lamivudine (300 mg), Zidovudine (300 mg), EPZICOM® (600 mg Ziagen® + 300 mg Lamivudine), COMBIVIR® (150 mg Lamivudine + 300 mg Zidovudine)
  The following NRTI combinations are prohibited in this study:
  * Didanosine + Stavudine
  * Zidovudine + Stavudine
  * Lamivudine + Emtricitabine

SUMMARY:
The purpose of this study is to determine the proportion of subjects with HIV-1 RNA < 50 c/mL at Week 48 in patients who failed their first line therapy containing a non-nucleoside reverse transcriptase inhibitor (NNRTI) or an integrase inhibitor

DETAILED DESCRIPTION:
Allocation: Randomization will be stratified

* ATV = Atazanavir
* DRV = Darunavir
* RTV = Ritonavir

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent.
* HIV-1 infected patients with viremia (VL ≥ 500/mL) on or after their first NNRTI or INI-based cART regimen and meeting one of the two criteria below:.

  i) On 1st line Non-nucleoside reverse transcriptase inhibitor (NNRTI) or Integrase inhibitor (INI)-based Combination antiretroviral therapy (cART) with HIV-1 RNA ≥ 500 c/ML after being on the same therapy for at least 12 weeks.

ii) Off 1st line NNRTI or INI-based Combination antiretroviral therapy (cART) for at least 2 weeks after having been on antiviral therapy for at least 4 weeks and who are non-compliant and off first line cART without a history of virologic failure with resistance, with a : HIV-1 RNA ≥ 500 c/ML.

* Fully sensitive genotype and phenotype report for Atazanavir/Ritonavir (clinical cut-off of 5.2) and Darunavir/Ritonavir (clinical cut-off ranging from 10 to 90).
* At least one NRTI other than Lamivudine (3TC) or emtricitabine (FTC) with full sensitivity (one "active" NRTI) by genotype and phenotype, ie, PhenoSense Genotype (GT), report must provide a "sensitive" net assessment of susceptibility. An NRTI or PI (reported with or without ritonavir) with a "partially sensitive" net assessment will not be considered "fully sensitive".
* Mentally able to participate in the study.
* Men and women ≥ 18 years old.
* Women of child bearing potential who engage in vaginal intercourse and who are not clinically sterilized must use highly effective methods of birth control during the study.

Exclusion Criteria

- Screening HIV genotype showing presence at baseline of any of the following Protease inhibitor (PI) Mutation Patterns associated with genotypic resistance to Atazanavir sulfate/ Ritonavir or Darunavir/Ritonavir will lead to exclusion:.

i) Subjects with any darunavir associated mutations* at baseline (*V11I, V32I, L33F, I47V, I50V, I54L, I54M, T74P, L76V, I84V and L89V).

ii) Subjects with a major mutation to Atazanavir sulfate consisting of N88S.

iii) Subjects with more than 3 of any of the following Atazanavir sulfate related mutations:D30N, M36I/V, M46I/L/T, I54V/L/T/M/A, A71V/T/I/G, G73S/A/C/T, V77I, V82A/F/T/S/I, I84V/A, N88D or L90M.

- Subjects with < 1 fully active NRTI on PhenoSense report, other than lamivudine and emtricitabine.

* Diagnosed with active tuberculosis.
* Chronic hepatitis B infection.
* Hepatitis C-positive patients who are not clinically stable or need treatment during the study period.
* Acute hepatitis in the 30 days prior to study entry.
* Any gastrointestinal disease or surgical procedure that may impact the absorption of study drug.
* Intractable diarrhea within 30 days prior to study entry.
* Presence of a newly diagnosed Human immunodeficiency virus (HIV)-related opportunistic infection or any medical condition requiring acute therapy at the time of enrollment.
* Subject's with Cushing's syndrome.
* Untreated hypothyroidism or hyperthyroidism.
* Recent therapy with agents with significant systemic myelosuppressive, neurotoxic, pancreatotoxic, hepatotoxic or cytotoxic potential within 3 months of study start.
* Subject's with obstructive liver disease.
* Active alcohol or illegal substance use.
* Inability to swallow capsules.
* Active peripheral neuropathy.
* Presence of cardiomypathy or any significant cardiovascular disease.
* Known, clinically significant cardiac conduction system disease.
* Physical and Laboratory Test Findings:.

  i) Moderate to severe hepatic insufficiency.

ii) Screening laboratory values as follows:.

A. T4 < 4mcg/dL or >11mcg/dL and/or Thyroid-stimulating hormone (TSH) <0.5mU/L or >5.0mU/L.

B. Calculated creatinine clearance < 60 cc/min.

C. Hemoglobin < 8.0 g/dL.

D. Total serum lipase ≥ 1.4 times the upper limit of normal (ULN).

E. Liver enzymes [Aspartate transaminase (AST), Alanine transaminase (ALT)] ≥ 5 times the ULN.

F. Alkaline phosphatase > 5 times the ULN.

G. Platelets < 50,000 cells/mm3.

H. Positive blood screen for hepatitis B surface antigen (HBsAg).

I. Total serum bilirubin ≥ 1.5 times the ULN.

- Allergies and Adverse Drug Reaction:.

i) Previously demonstrated hypersensitivity to any of the components of atazanavir or the other experimental agents in this study.

ii) Darunavir contains a sulfonamide moiety. Darunavir should be used with caution in patients with a known sulfonamide allergy.

iii) History of allergy to atazanavir, ritonavir, or darunavir.

iv) History of allergy to NRTIs included as NRTI backbone options in this study.

v) History of clinically relevant severe drug reaction.

- Sex and Reproductive Status:.

i) Women with a positive pregnancy test on enrollment prior to study drug administration.

ii) Women who become pregnant during the study will be taken off-protocol.

iii) Women using a prohibited contraceptive method.

iv) Women who are breastfeeding.

- Other Exclusion Criteria.

i) Prisoners or subjects who are involuntarily incarcerated.

ii) Subjects who are compulsorily detained for treatment of wither a psychiatric or physical illness.

- Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06-30 (Actual); Primary Completion 2014-08-31 (Estimated); Study Completion 2014-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with Human immunodeficiency virus 1 (HIV-1) Ribonucleic Acid (RNA) < 50 c/mL | At Week 48

SECONDARY OUTCOMES:
Proportion of subjects with HIV-1 RNA < 50 c/mL | At week 24
Change from baseline in CD4 cell count | Baseline (Week 0) and at week 48
Incidence rates of serious adverse event (SAEs) and adverse events (AEs) leading to discontinuation | up to week 48
Incidence rates of antiretroviral resistance measured by newly emergent genotypic substitutions and phenotypic resistance to study drugs for virologic failure | up to week 48
Proportion of subjects with HIV-1 RNA < 50 c/mL at Week 48 by baseline M184V presence or absence | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- United States (12):
  - Southwest Center For Hiv/Aids, Phoenix, Arizona
  - Health For Life Clinic Pllc, Little Rock, Arkansas
  - Anthony M. Mills Md Inc, Los Angeles, California
  - Uc Davis Medical Center, Sacramento, California
  - Metropolis Medical Pc, San Francisco, California
  - Indiana University Hospital, Indianapolis, Indiana
  - Be Well Medical Center, Berkley, Michigan
  - Southampton Health Center, St Louis, Missouri
  - I.D. Care Associates, Hillsborough, New Jersey
  - Saint Michael'S Medical Center, Newark, New Jersey
  - James J Peters VAMC, The Bronx, New York
  - Infectious Disease Clinic & AI, The Bronx, New York

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx